CLINICAL TRIAL: NCT02195505
Title: Use of Synvisc® in Knee Osteoarthritis - Medico-economical Study (U.S.A.G.E. Médico-Economique)
Brief Title: Use of Synvisc® in Knee Osteoarthritis - Medico-economical Study
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1139.1
Record Dates: First submitted 2014-07-18; First posted 2014-07-21 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2014-07

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Synvisc®
- Usual treatment of knee: nonsteroidal antiinflammatory drugs, antalgics

SUMMARY:
The USAGE study aims at assessing on a long-term period (two years in average) the outcome in clinical or economical term of patients with knee osteoarthritis (OA) treated or not with Synvisc®, in the 1139.4 clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients have already been followed up on a nine-month period in a pragmatic medica-economical clinical trial (BI Trial No.: 1139.4)

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: rheumatological practice
Sampling Method: Non-Probability Sample
Enrollment: 374 (Actual)
Dates: Start 2001-09; Primary Completion 2002-04 (Actual)

PRIMARY OUTCOMES:
Change in Lequesne index | up to 2 years
  assessment of algo-functional severity of pathology
Change in Womac index | up to 2 years
  assessment of symptom severity

SECONDARY OUTCOMES:
Medical costs related to knee osteoarthritis | up to 2 years